CLINICAL TRIAL: NCT04612933
Title: Effectiveness of Video Consultations in Type 1 Diabetes Patients Treated With Insulin Pumps in the Outpatient Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHS-MS-09-2020
Record Dates: First submitted 2020-10-15; First posted 2020-11-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Telemedicine; Insulin Dependent Diabetes Mellitus 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group video consultations (Experimental): All appointments, scheduled and non-scheduled are by telemedicine using video to commutate with the health care professionals.
  Patients will follow their usual treatment.
  Interventions: Other: Intervention group video consultations
- No intervention (No Intervention): All appointments, scheduled and non-scheduled are by face-face communication with the health care professionals.
  Patients will receive their usual treatment.

INTERVENTIONS:
Other: Intervention group video consultations — All appointments, scheduled and non-scheduled are by telemedicine using video to commutate with the health care professionals.
  Patients will follow their usual treatment.
  Arms: Intervention group video consultations

SUMMARY:
Telemedicine is a solution to overcome distance and ensure the provision of healthcare services. This study aims to investigate the effects of conducting outpatient clinic visits remotely, for patients living with insulin pumps.

DETAILED DESCRIPTION:
Telemedicine also has the potential to be a cost-effective solution due to reductions in travelling costs and saved working days, as well as increased patient satisfaction due to the reduction in transportation time.

Several studies have evaluated telemedicine for use in Diabetes Mellitus patients with an insulin pump. In all of these studies, the telemedicine group scheduled more contacts with the health care professionals than in the standard care group. To the investigator's knowledge, no one has investigated telemedicine, compared to standard care with the same number of scheduled contacts. The investigators believe telemedicine should increase the level of service and not increase the workload for health care professionals. A telemedical solution can provide patients with a more flexible alternative for visiting their health care provider rather having the burden of extra telemedicine appointments plus regular treatment.

Patients in rural Denmark may have a travelling time of 70 km (1 hour by car or several hours by public transport) to a specialised Diabetes Mellitus specialist centre. This may result in some patients choosing not to start or not being offered insulin pump treatment despite indications that an insulin pump is an optimal treatment choice. The challenge of distance also poses problems for patients in relation to technical problems or medical issues with the insulin pump. Telemedicine should be a solution for both patients and their Health Care Providers.

In this randomised controlled study, the effects of conducting clinical visits remotely, for patients living with insulin pumps will be investigated. Participants will be allocated to either Intervention (Standard care provide by video consultations) or standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age
* Diagnosed with diabetes Type 1
* Patient has used insulin pump for at least 6 months

Exclusion Criteria:

* No internet access
* Unable to adhere to protocol.
* Unable to speak or read Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Time in Range (TiR) | 52 weeks
  % of TiR (3.9 -10.0 mmol/L)

SECONDARY OUTCOMES:
Change from baseline of Glycaemic variability | 52 weeks
  (%GCV)
Change from baseline of Haemoglobin 1Ac | 52 weeks
  HbA1C %
Audit of Diabetes Dependent Quality of Life version 19 | 0 and 52 weeks
  Audit of Diabetes Dependent Quality of Life version 19 (ADDQoL 19) includes19 items each score from -9 to 3, with lower scores reflecting maximum negative impact.
Diabetes Treatment Satisfaction status | 0 and 52 weeks
  Diabetes treatment questionnaire, status (DTSQs) includes 8 items, each score from 0 to 6 with a higher score indicating better outcome
Diabetes Treatment Satisfaction Questionaire change | 52 weeks
  Diabetes treatment questionnaire, change (DTSQc) includes 8 items, each score from 3+ to -3 with a higher score indicating better outcome DTSQc
Change from baseline of time above target glucose range (TaR) level 1 | 52 weeks
  % TaR (10.1-13.9 mmol/L)
Change from baseline of time above target glucose range (TaR) level 2 | 52 weeks
  % TaR (>13.9 mmol/L)
Change from baseline of time spent below target glucose range (TbR ) level 1 | 52 weeks
  %TbR (3.0-3.8 mmol/L)
Change from baseline of time spent below target glucose range (TbR) level 2 | 52 weeks
  % TbR (<3.0 mmol/L)

OTHER OUTCOMES:
Changes in Quality of Life: EuroQol 5-Dimension 5-Level (EQ-5D-5L) | 0 and 52 weeks
  EQ-5D-5L includes 5 domains each score from 1 to 5 with level 1 indicating no problem and level 5 indicating unable to/extreme problems.
Semi-structured interviews | 0 and 52 weeks
  intervention group and Healthcare professionals

CONTACTS AND LOCATIONS:
Overall Officials: Frans Brandt Kristensen, MD, Ph.D., Study Director — Department of Endocrinology, Hospital of Southern Jutland
Locations (1):
- Sygehus Soenderjylland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang PH, Lau J, Chalmers TC. Meta-analysis of effects of intensive blood-glucose control on late complications of type I diabetes. Lancet. 1993 May 22;341(8856):1306-9. doi: 10.1016/0140-6736(93)90816-y. PMID 8098449
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Papatheodorou K, Papanas N, Banach M, Papazoglou D, Edmonds M. Complications of Diabetes 2016. J Diabetes Res. 2016;2016:6989453. doi: 10.1155/2016/6989453. Epub 2016 Oct 16. No abstract available. PMID 27822482
- [Background] Kannel WB, McGee DL. Diabetes and cardiovascular disease. The Framingham study. JAMA. 1979 May 11;241(19):2035-8. doi: 10.1001/jama.241.19.2035. PMID 430798
- [Background] Haffner SM, Lehto S, Ronnemaa T, Pyorala K, Laakso M. Mortality from coronary heart disease in subjects with type 2 diabetes and in nondiabetic subjects with and without prior myocardial infarction. N Engl J Med. 1998 Jul 23;339(4):229-34. doi: 10.1056/NEJM199807233390404. PMID 9673301
- [Background] Khoury JC, Kleindorfer D, Alwell K, Moomaw CJ, Woo D, Adeoye O, Flaherty ML, Khatri P, Ferioli S, Broderick JP, Kissela BM. Diabetes mellitus: a risk factor for ischemic stroke in a large biracial population. Stroke. 2013 Jun;44(6):1500-4. doi: 10.1161/STROKEAHA.113.001318. Epub 2013 Apr 25. PMID 23619130
- [Background] Laing SP, Swerdlow AJ, Carpenter LM, Slater SD, Burden AC, Botha JL, Morris AD, Waugh NR, Gatling W, Gale EA, Patterson CC, Qiao Z, Keen H. Mortality from cerebrovascular disease in a cohort of 23 000 patients with insulin-treated diabetes. Stroke. 2003 Feb;34(2):418-21. doi: 10.1161/01.str.0000053843.03997.35. PMID 12574553
- [Background] Stamler J, Vaccaro O, Neaton JD, Wentworth D. Diabetes, other risk factors, and 12-yr cardiovascular mortality for men screened in the Multiple Risk Factor Intervention Trial. Diabetes Care. 1993 Feb;16(2):434-44. doi: 10.2337/diacare.16.2.434. PMID 8432214
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Gaede P, Vedel P, Larsen N, Jensen GV, Parving HH, Pedersen O. Multifactorial intervention and cardiovascular disease in patients with type 2 diabetes. N Engl J Med. 2003 Jan 30;348(5):383-93. doi: 10.1056/NEJMoa021778. PMID 12556541
- [Background] Levin K, Madsen JR, Petersen I, Wanscher CE, Hangaard J. Telemedicine diabetes consultations are cost-effective, and effects on essential diabetes treatment parameters are similar to conventional treatment: 7-year results from the Svendborg Telemedicine Diabetes Project. J Diabetes Sci Technol. 2013 May 1;7(3):587-95. doi: 10.1177/193229681300700302. PMID 23759390
- [Background] Lee SWH, Ooi L, Lai YK. Telemedicine for the Management of Glycemic Control and Clinical Outcomes of Type 1 Diabetes Mellitus: A Systematic Review and Meta-Analysis of Randomized Controlled Studies. Front Pharmacol. 2017 May 30;8:330. doi: 10.3389/fphar.2017.00330. eCollection 2017. PMID 28611672
- [Background] Sood A, Watts SA, Johnson JK, Hirth S, Aron DC. Telemedicine consultation for patients with diabetes mellitus: a cluster randomised controlled trial. J Telemed Telecare. 2018 Jul;24(6):385-391. doi: 10.1177/1357633X17704346. Epub 2017 Apr 13. PMID 28406066
- [Background] Gonzalez-Molero I, Dominguez-Lopez M, Guerrero M, Carreira M, Caballero F, Rubio-Martin E, Linares F, Cardona I, Anarte MT, de Adana MS, Soriguer F. Use of telemedicine in subjects with type 1 diabetes equipped with an insulin pump and real-time continuous glucose monitoring. J Telemed Telecare. 2012 Sep;18(6):328-32. doi: 10.1258/jtt.2012.120103. Epub 2012 Aug 21. PMID 22912487
- [Background] Yaron M, Sher B, Sorek D, Shomer M, Levek N, Schiller T, Gaspar M, Frumkin Ben-David R, Mazor-Aronovitch K, Tish E, Shapira Y, Pinhas-Hamiel O. A randomized controlled trial comparing a telemedicine therapeutic intervention with routine care in adults with type 1 diabetes mellitus treated by insulin pumps. Acta Diabetol. 2019 Jun;56(6):667-673. doi: 10.1007/s00592-019-01300-1. Epub 2019 Feb 19. PMID 30783823
- [Background] Thomakos P, Mitrakou A, Kepaptsoglou O, Taraoune I, Barreto C, Zoupas CS. The Predictive Low Glucose Management System in Prevention of Clinically Significant Hypoglycemia in Type 1 Diabetes. A Preliminary Study Identifying the Most Common Events Leading Up to Hypoglycemia During Insulin Pump Therapy. Exp Clin Endocrinol Diabetes. 2021 May;129(5):385-389. doi: 10.1055/a-0889-7598. Epub 2019 Apr 15. PMID 30986882
- [Background] Rasmussen BS, Froekjaer J, Bjerregaard MR, Lauritsen J, Hangaard J, Henriksen CW, Halekoh U, Yderstraede KB. A Randomized Controlled Trial Comparing Telemedical and Standard Outpatient Monitoring of Diabetic Foot Ulcers. Diabetes Care. 2015 Sep;38(9):1723-9. doi: 10.2337/dc15-0332. Epub 2015 Jun 26. PMID 26116717
- [Derived] Schultz ANO, Christensen R, Bollig G, Kidholm K, Brandt F. Effectiveness of video consultations in type 1 diabetes patients treated with insulin pumps in the outpatient clinic: a randomised controlled trial. Diabetologia. 2026 Feb;69(2):321-329. doi: 10.1007/s00125-025-06585-2. Epub 2025 Nov 7. PMID 41198916
- [Derived] Schultz ANO, Christensen R, Bollig G, Kidholm K, Brandt F. Effectiveness of video consultations in type 1 diabetes patients treated with insulin pumps in the outpatient clinic: protocol for a randomised controlled trial. BMJ Open. 2022 Apr 27;12(4):e058728. doi: 10.1136/bmjopen-2021-058728. PMID 35477877